CLINICAL TRIAL: NCT03638791
Title: Longitudinal Study of Gut Microbiome in Obsessive-Compulsive Disorder
Brief Title: Microbiome in Obsessive-compulsive Disorder
Acronym: MIO
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Christian Rück, Head of Rucklab, affiliate professor, Karolinska Institutet
Other Study IDs: Microbiome in OCD
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Obsessive-Compulsive Disorder; Microbiota
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Biospecimen Retention: Samples With DNA — Stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy controls: Matched Controls without treatment
  Interventions: Behavioral: Exposure and response inhibition
- OCD: Exposure and response inhibition
  Interventions: Behavioral: Exposure and response inhibition

INTERVENTIONS:
Behavioral: Exposure and response inhibition — Cognitive behavioural therapy designed for treatment of Obsessive-compulsive disorder

SUMMARY:
Background: Humans live in symbiosis with microbes and their implication for health and disease is evident. The importance of microbiome-gut-brain axis in psychiatric disorders is an area of increasing research interest. OCD is a promising target for microbiome research as Pediatric Acute-onset Neuropsychiatric Syndrome (PANS)/ Pediatric autoimmune neuropsychiatric disorders associated with streptococcal infections (PANDAS) are reactions to infectious agents precipitating acute onset of severe OCD symptoms. Furthermore, preliminary evidence has associated probiotic treatment with alleviation of OCD symptoms. We propose the first clinical study on the microbiome and its effects on OCD patients.

Aim: To analyze the gut microbiota in patients with OCD compared with healthy matched controls and assess changes in microbial composition following treatment.

Outcome measures: Differences in alpha diversity, beta diversity, and taxa abundance of bacterial groups (at the phylum, class, order, family, genus and species levels) and severity of OCD symptoms. Moreover, functional profiling will be conducted.

Methods: Our aim is to enroll 32 OCD patients and 32 matched controls. Shotgun metagenomic sequencing will be used. Sequenced data will be processed followed by non-parametric statistical testing.

Significance: gut microbiome in patients with OCD beofre and after ERP treatment has never been done before. The microbial composition may impact on OCD symptoms, severity, and chronicity and could inform future therapeutic possibilities.

DETAILED DESCRIPTION:
Background:

Obsessive-compulsive disorder (OCD) is a highly debilitating disorder with a lifetime prevalence of approximately 2% is equally distributed among men and women. OCD generally starts at an early age and usually develops a chronic course if left untreated. Many patients with OCD receive treatment after years of delay due to both patient and health care factors; therefore, OCD affects educational achievement, ability to work and interpersonal relationships. Moreover, it poses a considerable burden and distress to family caregivers [1], and accounts for one of the ten most disabling mental health conditions worldwide [2].

The role of the microbial community in health and disease has been a neglected subject in human research until recently, despite the fact that human microbes comprise about 1-3 % of our body mass [3]. Gut microbes play important roles in nutrient metabolism, production of vitamins, and prevention of pathogens from colonizing our intestine [4]. Recently, microbiota in the gut has gained increasing interest due the extensive connection between the gut and the brain [5]. The bidirectional communication through neural, hormonal, and immunological signaling involving the central, autonomic, and enteric nervous systems forms the microbiome-gut-brain axis [6]. In psychiatry, dysbioses have been reported in anorexia nervosa, major depression, autism, and other major psychiatric disorders [9, 10].

Association between OCD onset and infection has long been known. PANS/PANDAS are acute-onset forms of OCD associated with autoimmune reactions from pathogens such as streptococcus infection [11, 12]. The connection between bacterial pathogen and immunological response, which generates OCD symptoms, is further evidence for the importance of the microbiome-gut-brain axis in OCD. Lately, there have been numerous hypotheses regarding the importance of gut microbiome and OCD symptoms [13, 14].

Aims: Characterize composition and diversity of the gut microbiome in individuals with OCD compared with healthy controls.

* We hypothesize that patients with OCD will show evidence of gut dysbiosis (imbalance) marked by lower microbial diversity and specific taxonomic and gene content differences compared to healthy controls. Primary outcome is α-diversity, which refers to the number of species (richness) at one site, β-diversity, which refers to the differences in species composition between participants, and taxonomic abundance of bacterial groups (at the phylum, class, order, family, genus, and species levels). These measures yield information about individual microbial composition at each site and homogeneity in a group of people.
* We hypothesize that reduced α and β diversity in gut microbiome correlate with severity of obsessive-compulsive symptoms measured by Yale-Brown Obsessive-Compulsive Scale (Y-BOCS), and Obsessive-Compulsive Inventory Revised (OCI-R). We predict that greater symptom severity is associated with lower diversity. A significant negative correlation will be supportive evidence for the microbiome-gut-brain axis.
* We hypothesize that there will be significant richer α diversity in gut microbiome composition after successful psychotherapy (change in Y-BOCS score).

Method:

Recruitment: Healthy controls will be recruited through advertisement or included from previous studies with their consent. Male and female patients between 18-45 years of age from the OCD-clinic at Huddinge Hospital with a DSM-5 diagnosis of OCD and fear of contamination will be invited to participate. Age matched controls will be recruited who have no personal or family history of OCD. Exclusion criteria for all groups include history of GI tract surgery (other than appendectomy or cholecystectomy); history of inflammatory bowel disease, irritable bowel syndrome, celiac disease, or any other diagnosis that could explain chronic or recurring bowel symptoms, antibiotic use in the past 3 months; pro-biotic use in the past 4 weeks; pregnantcy. Intellectual disability, autism spectrum disorder and psychosis.

Assessment: All participants will meet an experienced psychiatrist for diagnostic assessments including M.I.N.I. interview. Participants will be asked to complete self-assessment forms on the Internet and answer questions about their dietary habits for the last three months. Weight and height for body mass index (BMI) calculation will be measured. All assessment forms, information from interviews and medical examination will be documented in their medical record. Further information (e.g. antibiotics and previous therapies) will be collected from their medical records with the participants' consent.

The investigators chose the following questionnaire battery to capture all relevant outcome variables (OCD-symptoms), nutrition, and stool characteristics and frequency.

* Yale-Brown Obsessive Compulsive Scale (Y-BOCS): A commonly used clinical, semi-structured interview assessing severity of OCD symptoms.
* Obsessive-Compulsive Inventory Revised (OCI-R -): An18 item self-report questionnaire estimating OCD symptom dimensions.The OCI-R yields a total score and 5 subscales: checking, hoarding, neutralizing, obsessing, ordering and washing.
* EDE-Q to capture eating behavior.
* Meal Q questionnaire: A web-based food frequency questionnaire normed in Sweden will validate energy and macronutrient intake, which affects the microbial composition.
* Bristol Stool Scale: A medical diagnostic scale designed to classify the form of human faeces into seven categories.

Furthermore, the investigators will collect demographic information of all patients: age, sex, age at onset, occupation status, somatic health, and psychiatric comorbidities.

Stool sampling procedure: Patients and controls will be provided with clear instructions for home fecal sample collection. Patients will collect one stool sample at the beginning of treatment and one at the end of treatment. Controls will collect one sample at one time point only. Participants will collect stool at home using OMNIgene kits that will be sent to the KI biobank.

Exposure and Respons Prevention therapy (ERP): an evidence-based psychotherapy administered by experienced psychologists, either individually, in groups, face-to-face or through internet. A minimum of five exposure and respons prevention sessions is required in order for it to be considered an ERP treatment.

Sample storage in biobank: All samples will be stored at Karolinska Institutets (KI) biobank. Application for biobank storage of samples is established according to rules and regulations.

Metagenomic sequencing: The investigators will use shotgun metagenomics sequencing methods. Whole-genome shotgun sequencing can provide functional information on which genes are present in the gut microbiome of patients. This method can also provide a more detailed taxonomical resolution that 16S rRNA sequencing.

Metagenomic shotgun sequencing: will be prepared and sequenced. To efficiently utilize the flow cells, about ten samples will be multiplexed, with dual indices, per lane of the flow cell. Prior to downstream bioinformatics analysis, raw sequence data will be quality filtered and trimmed to remove bases with Phred quality scores less than 20. Data generated will be processed by metagenome species concept. Sequences are clustered into metagenomic species (MGS) based on their sequence similarity.

Determination of sample size: two previous studies with fewer or similar number of participants have shown that this study will be adequately powered. Furthermore, this is a pilot study based on new sequencing technology.

Timeline: Ethical application has been approved and all samples have been collected.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of OCD. Age matched controls will be recruited who have no personal or family history of OCD.

Exclusion Criteria:

* history of GI tract surgery (other than appendectomy or cholecystectomy); history of inflammatory bowel disease, irritable bowel syndrome, celiac disease, or any other diagnosis that could explain chronic or recurring bowel symptoms, antibiotic use in the past 3 months; pro-biotic use in the past 4 weeks; pregnancy. Intellectual disability, autism spectrum disorder and psychotic disorders.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Recruitment of participants from Karolinska Hospital in Solna and Huddinge. Healthy Controls are recruited from Sweden from advertisements.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2022-09-04 (Actual); Study Completion 2022-09-04 (Actual)

PRIMARY OUTCOMES:
Alpha diversity | 2018-09-01
  expressed as number of observed species and Chao-1 estimator

SECONDARY OUTCOMES:
Beta diversity | 2018-09-01
  UniFrac distances
Taxonomic and functional differences between cases and controls | 2018-09-01
  Metagenomic species and gut-brain modules
Change in microtioba diversity before and after ERP treatment | 2018-09-01
  Change in alpha diversity before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christian Rück, MD, Study Chair — Karolinska Institutet; Diana Radu Djurfeldt, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- M46: Karolinska Universitetssjukhuset, Psykiatri Sydväst, Stockholm, Huddinge, Sweden